CLINICAL TRIAL: NCT04290013
Title: Effect of Tranexemic Acid and Norethisterone Acetate on Endometrial Vasculature in Women With Dysfunctional Uterine Bleeding.
Brief Title: Effects of Tranexemic Acid Versus Norethisterone Acetate on Endometrial Vasculature .
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Elkattan, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol 400
Record Dates: First submitted 2020-02-23; First posted 2020-02-28 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Dysfunctional Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Norethindrone Acetate; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- norethisterone -women with Dysfunctional uterine bleeding (Experimental)
  Interventions: Drug: norethisterone acetate
- tranexemic acid-women with Dysfunctional uterine bleeding (Experimental)
  Interventions: Drug: tranexamic acid tablets

INTERVENTIONS:
Drug: norethisterone acetate — norethisterone acetate 15 mg daily from day 5 of the cycle to day 26.
  Arms: norethisterone -women with Dysfunctional uterine bleeding
Drug: tranexamic acid tablets — tranexemic acid 1 gm three times daily from the first day of the menstrual cycle up to 5 days .The dose can be increased but not exceeding 4 gm per day.
  Arms: tranexemic acid-women with Dysfunctional uterine bleeding

SUMMARY:
Heavy periods is a significant problem in reproductive age .It affects about a third of women in the childbearing period

Any of the following is considered to be heavy menstrual bleeding (Bleeding that lasts more than 7 days,Bleeding that soaks through one or more tampons or pads every hour for several hours in a row.Needing to wear more than one pad at a time to control menstrual flow.,Needing to change pads or tampons during the night or Menstrual flow with blood clots that are as big as a quarter or larger) .

Heavy periods can be caused by organic cause as fibroids, adenomyosis, polyps or they can be dysfunctional.Dysfunctional uterine bleeding is irregular uterine bleeding that occurs in the absence of recognisable pelvic pathology, general medical disease, or pregnancy. It reflects a disruption in the normal cyclic pattern of ovulatory hormonal stimulation to the endometrial lining.

Several treatment options include: hormonal treatment as norethisterone acetate,oral contraceptive pills, gonadotrophin releasing hormone analogue. ,tranexamic acid or non steroidal anti-inflammatory drugs.

The investigators plan to do a comparative study between norethisterone acetate and tranexamic acid regarding their control of the heavy periods as well as their effect on the uterine and endometrial vasculature.

DETAILED DESCRIPTION:
This is a Randomised controlled trial.The investigators will randomise 120 women who suffer from heavy periods (age range 35-49 years old) without organic cause (Dysfunctional bleeding ) into 2 groups, group A (60 women) : They will take norethisterone acetate 15 mg daily from day 5 to day 26 of the period for 3 months.

Group B (60 women): They will take 1 gm tranexemic acid three times daily from the start of menstrual period up to 5 days.The dose might be increased per day (Not more than 4 gm per day).

The investigators will check endometrial thickness, endometrial volume, uterine artery Doppler indices as well as endometrial and subendometrial indices before starting the treatment and 3 months afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Age: 35-49 years old.
* Normal gynecologic and breast examination
* Women who have sterilization or husband is sterilized or accepts to use a suitable barrier contraception during the duration of the study.
* Heavy periods (were assessed by validated pictorial blood chart)
* Normal ultrasound, hysteroscopy and endometrial biopsy.
* Normal coagulation profile and thyroid function.
* No contraindication to tranexamic acid or Norethisterone acetate : allergy,History of arterial or venous thromboembolic disease,Disturbance of liver function or Severe renal impairment.

Exclusion Criteria:

* Women who are less than 35 years old or more than 49 years old.
* Women who had organic cause for heavy periods as uterine polypi,fibroids or endometriosis.
* Women taking hormonal preparation the month before starting the trial.
* Women with abnormal findings in pelvic ultrasound,hysteroscopy or endometrial biopsy.
* Women who suffer from uncontrolled diabetes or uncontrolled hypertension.
* Women with history of breast cancer or precancerous conditions.

Ages: 35 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2020-04-22 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
reducion of the menstrual flow. | 3 months
  Using Pictorial Blood loss assessment chart depends on counting the sanitary pads and scoring the amount of blood in them)

SECONDARY OUTCOMES:
endometrial thickness in centimetre. | Before the intervention and 3 months afterwards
  Measurement of the thickest part of the endometrium in centimetres in the longitudinal plan of the uterus using Two- Dimensional Transvaginal ultrasound
endometrial volume in cubic centimetre. | Before the intervention and 3 months afterwards
  Measurement of the endometrial volume in cubic centimetres using Three-Dimensional transvaginal ultrasound
uterine artery Doppler indices. | Before the intervention and 3 months afterwards
  Measurement of the uterine artery Doppler indices using Transvaginal ultrasound and taking the mean for both arteries.
endometrial three-dimensional vascular indices. | Before the intervention and 3 months afterwards
  Measuring the vascularity in the endometrium using power doppler and Three -Dimensional transvaginal ultrasound.

IPD SHARING:
Plan to Share IPD: Undecided